CLINICAL TRIAL: NCT05491434
Title: Intervention, Non-randomized Controlled, Non-masked and Comparative Study of Presurgical Conditioning in Colorectal Cancer Patients Who Present With Sarcopenia
Brief Title: Sarcopenia in Colorectal Cancer Patients, Intervention Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, Ricardo Frago Montanuy, PhD, Hospital Universitari de Bellvitge
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: PR137/19
Record Dates: First submitted 2022-08-04; First posted 2022-08-08 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Sarcopenia; Postoperative Complications; Infection;Post Surg Procedure
Keywords: Sarcopenia; Colon cancer; Postoperative complications; Inmunologic status; L3 CT image
MeSH Terms: conditions — Sarcopenia; Postoperative Complications; Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): The usual pre-surgical preparation and conditioning will be carried out, without providing nutritional supplements or increased physical activity
- Experimental (Experimental): In addition to the usual pre-surgical preparation and conditioning, a nutritional supplement and increased physical activity will be provided in a controlled manner for 3 weeks.
  Interventions: Dietary Supplement: Protein supplement

INTERVENTIONS:
Dietary Supplement: Protein supplement — One líquid brick every day during 3 weeks
  Other Names: 10gr protein/100 ml. Every liquid brick have 200 ml
  Arms: Experimental

SUMMARY:
The sarcopenia is a new concept for evaluating the functional status of patients, introduced during the last 20 years. This is defined as the relationship between the deterioration of muscle mass and the decrease in strength, the metabolic rate, the aerobic capacity and subsequently the evaluation of the functional status. The sarcopenia has been estimated to affect 5% to 13% of people aged between 60 and 70 years, increasing from 11% to 50% in those aged 80 years and older. In a study by Lieffers et al. of a total of 234 patients with colorectal cancer, with a mean age of 63 years according to the values observed by Prado et al., the prevalence of sarcopenia would be around 39%, being able to reach up to 60% in patients with chronic diseases.

The goal of this study is to compare the cumulative incidence of post-surgical complications due to infection at 30 days between the group of patients without sarcopenia and the group of patients with sarcopenia with an intervention based on a nutritional supplement + physical exercise.

DETAILED DESCRIPTION:
CONCEPTUAL HYPOTHESIS Improving functional status through physical exercise and nutritional supplementation of sarcopenic colon cancer patients at diagnosis can reduce the rate of infectious complications after surgery.

OPERATIONAL HYPOTHESIS Active preoperative preparation of sarcopenic colon cancer patients reduces post-surgical infectious complications by at least 11%, reaching a rate similar to patients without initial sarcopenia.

Inclusion criteria: - Age ≥ 70 years old; - Colon adenocarcinoma without synchronous metastases; - No urgent surgery; - ECOG performance status ≤ 2 .; - no pregnancy or lactation .; - signature of the informed consent; - ability to comply with the study indications. Exclusion criteria: - rectal cancer; - Concomitant neoplastic disease in the last 5 years - medical or mental condition of the patient that compromises the authorization of informed consent; - Concomitant uncontrolled or stable medical condition; - Clinically significant heart disease (congestive heart failure, symptomatic coronary disease) - Refusal to participate in the study.

Study variable (categorization of patients): Evaluation of Sarcopenia: it will be performed by CT, identifying the image of L3 (3rd lumbar vertebra). Main outcome variable: Cumulative incidence of post-surgical complications due to infection at 30 days.

Secondary variables: Frailty, Immune status, Quality of life (QoL) C30 and CR29 INTRVENTION (study groups)

* ARM A (Control: No sarcopenia): the usual pre-surgical preparation and conditioning will be carried out, without providing nutritional supplements or increased physical activity.
* ARM B (Experimental: Sarcopenia): in addition to the usual pre-surgical preparation and conditioning, a nutritional supplement and increased physical activity will be provided in a controlled manner for 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 70 years old,
* Colon adenocarcinoma without synchronous metàstasis,
* No urgent surgery,
* ECOG performance status ≤ 2,
* no pregnancy or lactation,
* signature of the informed consent,
* ability to comply with the study indications.

Exclusion Criteria:

* rectal càncer,
* Concomitant neoplastic disease in the last 5 years
* medical or mental condition of the patient that compromises the authorization of informed consent,
* Concomitant uncontrolled or stable medical condition,
* Clinically significant heart disease (congestive heart failure, symptomatic coronary disease)
* Refusal to participate in the study.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 370 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
to evaluate the rate of post-surgical infectious complications between the group of sarcopenic and non-sarcopenic patients | 30 days
  Evaluate the cumulative incidence of post-surgical complications due to infection at 30 days between the group of patients without sarcopenia and the group of patients with sarcopenia with an intervention based on a nutritional supplement + physical exercise in the latter group

SECONDARY OUTCOMES:
To asess the rate of post-surgical complications between the group of sarcopenic and non-sarcopenic patients | 30 days
  All complications, not just infectious
Overall survival at one year | One year
  To study survival one year after surgery in patients considered preoperatively as having sarcopenia.
Quality of life of surgical patients | At 3 months, 6 months and one year after surgery
  Evaluate the quality of life according the QLQ EORTC QlQ C-30 y ClQ CR29

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain